CLINICAL TRIAL: NCT06924541
Title: Choline Dose Ranging and Brain Functioning in Postmenopausal Women
Brief Title: Choline Dose Ranging in Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Dumas (Other)
Responsible Party: Sponsor-Investigator, Julie Dumas, Professor, University of Vermont
Organization: University of Vermont (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STU3122
Record Dates: First submitted 2024-08-19; First posted 2025-04-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Menopause
Keywords: cognition; fMRI; working memory
MeSH Terms: interventions — Choline

STUDY DESIGN:
Intervention Model Description: Placebo controlled study
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Choline low 550 mg dose (Experimental): Each subject completes three study days with a low and higher dose of choline and placebo
  Interventions: Dietary Supplement: Choline
- Choline higher 1100 mg dose (Experimental): Each subject completes three study days with a low and higher dose of choline and placebo
  Interventions: Dietary Supplement: Choline
- Placebo (Placebo Comparator): Each subject completes three study days with a low and higher dose of choline and placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Choline — Each subject gets one of two oral choline doses or placebo on each of three study days, 550 mg, 1100 mg, and placebo
  Arms: Choline higher 1100 mg dose; Choline low 550 mg dose
Dietary Supplement: Placebo — Each subject gets one of two oral choline doses or placebo on each of three study days, 550 mg, 1100 mg, and placebo
  Arms: Placebo

SUMMARY:
This study will use a randomized placebo-controlled trial to examine smaller doses of choline and whether a signal in the brain is detectable using fMRI. This study will examine if an even smaller doses of choline can show these similar brain activation and connectivity patterns to the 1650 mg dose. This will be a dose ranging study of 550 mg and 1100 mg oral choline compared to placebo.

DETAILED DESCRIPTION:
The brain is a major target for circulating gonadal steroids and the change in hormone levels after menopause is likely to have implications for cognitive functioning. Clinical and preclinical studies have linked gonadal steroids and cognition and it has been hypothesized that menopause has detrimental effects on cognition that are over and above the expected effects of normal aging. However, evidence for changes in cognition after menopause is equivocal. Some studies found decreased cognitive performance after menopause in domains such as memory, attention, problem solving, and motor skills. Other studies have not found changes in cognition after menopause. Additionally, not all women experience negative effects of menopause on cognition. The neurobiological processes underlying individual differences in cognition after menopause are not fully understood.

Choline is an essential nutrient that, in addition to its role in the brain, has a number of critical structural and physiologic roles throughout the body, including providing structural integrity and signaling function for cell membranes, facilitating lipid transport from the liver, and acting as the major source of methyl groups through diet. Aside from dietary intake, the only source of choline in the body is de novo synthesis of phosphatidylcholine, catalyzed by phosphatdylethanolamine-N-methyltransferase (PEMT). The PEMT gene has several estrogen-responsive components in its promoter region and is induced by estrogen. Post-menopausal (hypo-estrogenic) women with loss of function mutations in PEMT have been found to exhibit end-organ damage typical of choline deficiency.

Choline is also involved in the synthesis of acetylcholine, a major neurotransmitter and the central and peripheral nervous systems. The relationship between brain effects of the normal functioning of the cholinergic system and hormone changes after menopause has been demonstrated in preclinical studies in rat models and in experimentally in human studies. While the preclinical and clinical experiment studies have many similar findings regarding the influence of estrogen on cholinergic functioning, what is not clear from this research is how individual differences arise in the effects of the hormone withdrawal after menopause on brain functioning in middle aged women. It is possible that the estrogen control of the transcription of the PEMT gene may influence the availability of choline.

The investigators recently completed a study of one oral dose of 1650 mg choline versus placebo in 20 healthy postmenopausal women aged 50-65 years. Choline or placebo was administered three hours before an MRI session where subjects underwent an MRS scan as well as functional MRI scans. The MRS scans did not show differences in choline levels in the brain between the choline and placebo study days. However, the functional MRI (fMRI) results showed that choline modulated activation patterns during working memory task as well as influenced functional connectivity between memory relevant regions in the brain. The pattern of activation showed that during the choline challenge compared to placebo, there was decreased frontal activation and increased posterior activation during working memory. The functional connectivity analysis showed decreased connectivity during choline compared to placebo. This pattern of activation is similar to what has been shown with estradiol administration in healthy postmenopausal women. Recent choline data and prior estrogen data resulted in brain activation patterns similar to those of younger adults when compared to older adults. These results were interpreted to indicate that choline in a similar way to estradiol resulted in more efficient patterns of brain activation in healthy postmenopausal women.

This study will use a randomized placebo-controlled trial to examine smaller doses of choline and to detect a signal in the brain using fMRI. This study will examine if even smaller doses of choline can show these similar brain activation and connectivity patterns to the 1650 mg dose. This is a dose ranging study of 550 mg and 1100 mg oral choline compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-65 years
* Postmenopausal: Women who are postmenopausal will have not had a period in the last 12 months, have FSH>30 IU/L, and estradiol (E2) <50 pg/ml.
* Nonsmokers
* Not taking hormone therapy, SSRIs, phytoestrogens, SERMS, or antiestrogen medications and will be at least one year without such treatment
* Physically healthy
* No cardiovascular disease other than mild hypertension. Subjects will also not have current untreated or unremitted Axis I or II psychiatric or cognitive disorders (see screening below).
* IQ in the normal range >80
* Normal neuropsychological test performance

Exclusion Criteria:

* MCI or dementia - Montreal Cognitive Assessment <26, Mattis Dementia Rating Scale <130, and Global Deterioration Scale >2
* History of cancer treatment with cytotoxic and/or ongoing (current) maintenance targeted chemotherapy
* Blood pressure > 160/100 (untreated)
* Untreated thyroid disease
* Significant cardiovascular disease
* Asthma or COPD
* Active peptic ulcer
* Hyperthyroidism
* Epilepsy
* Current untreated or unremitted Axis I psychiatric disorders Use of medications on the Prohibited medications (see list)

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
BOLD Signal during fMRI working memory task | measured on each of the three study days
  fMRI BOLD signal during a working memory task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided
After data are published, deidentified data will be made available to those who request access